CLINICAL TRIAL: NCT06648954
Title: Multisite High-definition Transcranial Direct Current Stimulation Targeting Sensorimotor Network Navigated by Task-based fMRI to Facilitate Motor Activation and Reorganization for Stroke
Brief Title: Effect of Multisite High-definition Transcranial Direct Current Stimulation Targeting Sensorimotor Network
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018.661b
Record Dates: First submitted 2024-09-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multisite HD-tDCS group (Experimental): Device:
  Constant current will be applied for 20min and the electrodes will be placed over the target area
  Interventions: Device: multisite HD-tDCS
- Sham stimulation group (Sham Comparator): The stimulator will be applied for 20 minutes with only 30s ramp-up and ramp-down stimulation delivered. The patients will feel the initial itching sensation at the beginning in order to evaluate the placebo effect.
  Interventions: Device: Sham stimulation
- Conventional tDCS Group (Active Comparator): Constant current (2mA) will be applied for 20min and the anode will be placed over the standard C3/C4 position.
  Interventions: Device: Conventional tDCS

INTERVENTIONS:
Device: multisite HD-tDCS — 5-8 MRI compatible electrodes (2 cm diameter) will be placed based on the neuroimaging and computation modelling. The electrodes will be placed inside MRI compatible sponges and affixed to the head using a device matched cap which will be filled with saline to have good contact with the scalp.
  Arms: Multisite HD-tDCS group
Device: Conventional tDCS — A pair of 25 cm2 rubber electrodes enclosed in saline-soaked sponges and affixed to the head with rubber bands.
  Arms: Conventional tDCS Group
Device: Sham stimulation — 5-8 MRI compatible electrodes (2 cm diameter) will be placed based on the neuroimaging and computation modelling. The electrodes will be placed inside MRI compatible sponges and affixed to the head using a device matched cap which will be filled with saline to have good contact with the scalp.
  Arms: Sham stimulation group

SUMMARY:
Transcranial direct current stimulation (tDCS) has been applied to facilitate cortical excitability in stroke populations, as increasing evidence suggests that clinical recovery from stroke is attributed to neuroplastic reorganization. However, recovery from stroke following this kind of non-invasive neuromodulation remains divergent across stroke patients due to variations in their etiologies, lesion profiles and post-stroke duration.

A novel multisite high definition tDCS (HD-tDCS) in healthy people showed that such network-targeted stimulation could enhance motor excitability beyond conventional stimulation which targeting only one region. The electrode placements could be determined by the montage optimization, which targets individual motor network activation navigated by task-based fMRI using computation algorithms.

By targeting motor network, the new multisite electrode montage may provide a potential to facilitate better cortical activation than conventional tDCS montage.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) has been applied to facilitate cortical excitability in stroke populations, as increasing evidence suggests that clinical recovery from stroke is attributed to neuroplastic reorganization. However, recovery from stroke following this kind of non-invasive neuromodulation remains divergent across stroke patients due to variations in their etiologies, lesion profiles and post-stroke durations. In the stroke application of tDCS, most non-invasive brain stimulation studies have mainly focused on the modulation of the primary motor cortex (M1) in motor skill relearning. Previous studies have shown that not only the M1, which is the most important area associated with the motor system, but also other secondary motor areas (e.g., premotor cortex (PM) and supplementary motor area (SMA)) can be influenced by the onset of stroke. In fact, SMA activations and shifts in the M1 are commonly observed in stroke patients. However, brain regions do not operate in isolation, but communicate and interact with other discrete regions through networks. Conventional stimulations of one region (normally the M1 in stroke) have neglected the network impact and the changed motor network composition after stroke, which is often limited in stroke rehabilitation. A novel multisite high definition tDCS (HD-tDCS) in healthy people showed that such network-targeted stimulation could enhance motor excitability beyond conventional stimulation which targeting only one region. It showed that the excitability following multisite HD-tDCS was more than double the increase following conventional tDCS.

To consider the various lesion site and the different activation patterns of individual stroke survivors, personalized lesion profiles and anatomical features can be determined using finite element modelling, with lesion profiles generated from MRI and advanced algorithms calculating the current density to maximize the modulation effect. The electrode placements could be determined by the montage optimization, which targets individual motor network activation navigated by task-based fMRI using computation algorithms. By targeting motor network, the new multisite electrode montage may provide a potential to facilitate better cortical activation than conventional tDCS montage.

In this study, A randomized cross-over designed trial will be conducted to explore motor activation and reorganization changes before and after multisite HD-tDCS, conventional tDCS, and sham tDCS in stroke survivors. The stimulation effect will be evaluated by fMRI.

ELIGIBILITY:
Inclusion Criteria:

1. first-ever stroke, the duration after stroke exceeds 12 months;
2. mild to moderate upper extremity motor function deficit, determined by the Fugl-meyer assessment of upper extremity (FMAUE) scores between 15 and 53;
3. could voluntarily perform grasping hand movement.
4. sufficient cognitive function to follow the assessment and experiment instructions.

Exclusion Criteria:

1. history of epilepsy, or any other contradictions of brain stimulation and MRI scanning;
2. severe joint contracture of elbow or shoulder, or pain induced by any other neurological, neuromuscular, and orthopedic diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting-state functional connectivity | before and immediately after stimulation
  Functional magnetic resonance imaging for collecting BOLD signals during resting-state.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | before experiment
  Motor function assessment for stroke survivors
task-based brain activation | before and immediately after stimulation
  Functional magnetic resonance imaging for collecting BOLD signals during motor tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kai-yu Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong